CLINICAL TRIAL: NCT02169596
Title: a Single Centre Open Pilot Study to Explore if the Efficacy of PLAtelet Aggregation Inhibition by Ticagrelor Mediated P2Y12 Blockade Dependent Upon Endogenous Endothelial Nitric OXide?
Brief Title: Is Efficacy of PLAtelet Aggregation Inhibition by Ticagrelor Mediated P2Y12 Blockade Dependent Upon Endogenous Endothelial Nitric OXide?
Acronym: PLATE NOX
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLATE NOX; 14/YH/0179 (Other: SouthYorks NRESCommittee.YorkandHumber- (HEALTH RESEARCH AUTHORITY))
Record Dates: First submitted 2014-06-17; First posted 2014-06-23 (Estimated); Last update posted 2019-07-15 (Actual); Status verified 2019-07

CONDITIONS: Acute Coronary Syndome
Keywords: Acute Coronary Syndrome; Nitric oxide; Ticagrelor; Antiplatelet agents; Endothelial function
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Ticagrelor; Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coronary Artery Disease (Other): Blood tests to assess platelet function and EndoPAT assessment for endothelial function testing before and after ticagrelor administration (90mg BD)
  Interventions: Drug: Ticagrelor; Other: EndoPAT - endothelial assessment
- Healthy Normals (Other): Blood tests to assess platelet function and EndoPAT assessment for endothelial function testing before and after ticagrelor administration (90mg BD)
  Interventions: Drug: Ticagrelor; Other: EndoPAT - endothelial assessment

INTERVENTIONS:
Drug: Ticagrelor — Blood tests taken for flow cytometry
  Other Names: blood test
Other: EndoPAT - endothelial assessment

SUMMARY:
Background

Acute coronary syndrome (ACS) is a term representing all diseases related to reduction in blood flow to the heart characterised by clot formation over a segment of blood vessel narrowing. A major constituent of clot are blood cells called platelets and many of the medications used in ACS target platelet function. Ticagrelor is known to reduce platelet activity in clot formation by blocking a specific step in the process (P2Y12 receptors). A recent study has found that the presence of ticagrelor may also reduce clot formation by significantly enhancing another process involving the molecule nitric oxide (NO). This is of particular interest if translates into clinical practice, as many patients with heart disease have abnormal function of their blood vessel lining. This is known to cause a reduction in available nitric oxide. Does this therefore mean these patients will have a reduced response to ticagrelor therapy and subsequently be at increased risk of clot formation?

Aims

1. Will ticagrelor increase the anti clot effect of vessel lining produced nitric oxide?
2. Do patients with diabetes or smokers, who have poor function of their vessel lining, have a reduced response to ticagrelor?

Methods

This is a pilot study in which we propose to look at 64 patients with known disease of their heart blood vessels, with an equal mix of smokers, diabetics, smoking diabetics and non smoking non diabetics. We will also recruit ten healthy normal subjects to ensure that our tests produce the same results as the basic science study mentioned above.

To answer the questions posed we will perform blood tests, primarily looking at platelet function, and non-invasive blood vessel lining assessment. This will be done before and after ticagrelor treatment on each participant, enabling statistical comparison.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Coronary artery disease deemed to require Percutaneous Coronary Intervention
* Diabetics must be established on oral or subcutaneous therapy
* Non diabetics must have HbA1c levels between 20-42 mmol/mol
* Current smokers are those that have smoked greater than 100 cigarettes and currently smoke on a daily basis
* Non smokers have not smoked for greater than 3 years (and not on nicotine replacement)
* Healthy controls are non smokers without medical history and taking no regular medication

Exclusion Criteria:

* Contra-indication to dual antiplatelet therapy

  * Known bleeding disorders
  * Known malignant disease
  * Known myeloproliferative disease/malignant paraproteinaemia/heparin induced thrombocytopenia
  * Previous intracranial bleed
* Already established on dual antiplatelet therapy
* Known moderate-severe liver or splenic failure
* Severe renal impairment
* Major surgery due within one month of enrolment or before completion of measurements
* Known allergy/intolerance to aspirin or ticagrelor
* Reaction or side effect of aspirin or ticagrelor resulting in discontinuation prior to completion
* Known allergy/intolerance to 3-hydroxy-3-methylglutaric acid Coenzyme A reductase inhibitor therapy (statins)
* Concurrent use of high dose simvastatin/lovastatin (>40mg daily)
* Currently taking medication that will interact with platelet function ie NSAIDS, antibiotics or herbal remedies
* Concurrent use of strong cytochrome P450 3A4 inhibitors eg. ketoconazole, clarithromycin, nefazodone, ritonavir, and atazanavir
* Concurrent use of strong cytochrome P450 3A4 inducers e.g. rifampicin, dexamethasone, phenytoin, carbamazepine and phenobarbital
* Known sick sinus syndrome, second or third degree AV block or bradycardia-related syncope without permanent pacemaker in situ
* Known severe asthma/Chronic Obstructive Pulmonary Disease or worsening of dyspnoeic symptoms on ticagrelor
* Known severe gout
* Currently taking calcium channel antagonist
* Currently taking long acting nitrate
* Currently taking >15mg/week of methotrexate
* Women pregnant, breast feeding or of child bearing potential
* Require anticoagulation on warfarin or Novel Oral AntiCoagulant
* Platelet count <150 x109/L or >400 x109/L
* Known blood bourne virus carrier
* Unable to give informed consent
* Involvement in a conflicting study
* Non English speaker

Withdrawal Criteria following initial recruitment due to not meeting inclusion or exclusion criteria

* Develop significant bleeding complications of medication requiring discontinuation of antiplatelet therapy prior to completion of the study
* Urgent surgery undertaken during the study resulting in discontinuation of antiplatelet therapy prior to completion of the study
* React or develop side effects of aspirin or ticagrelor resulting in discontinuation prior to completion of the study
* Commence medication that will interact with platelet function before completion of the study
* Commence use of strong cytochrome P450 3A4 inhibitors before completion of the study
* Commence use of strong cytochrome P450 3A4 inducers before completion of the study
* Worsening of dyspnoea in subjects with mild/moderate asthma/Chronic Obstructive Pulmonary Disease resulting in discontinuation of ticagrelor prior to completion of the study
* Platelet count on initial sampling <150 x109/L or >400 x109/L
* Non diabetic patients HbA1c level >42 mmol/mol
* Noncompliance with medication
* Subject wishes to no longer participate in the study (no reason or time period required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Platelet Function | up to 12 months (completion of study)
  Direct testing with flow cytometry measuring fibrinogen binding, P-selectin, CD40L expression

SECONDARY OUTCOMES:
Reactive Hyperaemia Index | at 1 month, 6 months and at 12 months (completion of study)
  EndoPAT endothelial assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Castle Hill Hospital (Hull and east Yorkshire Hospitals NHS Trust), Cottingham, East Yorkshire, United Kingdom

REFERENCES:
- [Result] Rossington JA, Brown OI, Hoye A. Systematic review and meta-analysis of optimal P2Y12 blockade in dual antiplatelet therapy for patients with diabetes with acute coronary syndrome. Open Heart. 2016 Feb 26;3(1):e000296. doi: 10.1136/openhrt-2015-000296. eCollection 2016. PMID 27127634
- See also: Publication Link — https://openheart.bmj.com/content/3/1/e000296